CLINICAL TRIAL: NCT00000815
Title: A Phase II, Comparative Study of Seroconversion of Single-Dose and Two-Dose Measles Vaccination in HIV-Infected and HIV-Uninfected Children: A Multicenter Trial of the Pediatric AIDS Clinical Trials Group
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG 225; 11202 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Measles
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Measles-Mumps-Rubella Vaccine; Vaccines, Attenuated; Measles Vaccine; Immunization Schedule; Measles Virus; Measles
MeSH Terms: conditions — HIV Infections; Measles; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Measles Vaccine; Measles-Mumps-Rubella Vaccine

ARMS (2):
- 1 (Experimental): Participants who receive vaccination at 6 and 12 months of age
  Interventions: Biological: Attenuvax; Biological: M-M-R-II
- 2 (Experimental): Participants who receive vaccination only at 12 months of age
  Interventions: Biological: M-M-R-II

INTERVENTIONS:
Biological: Attenuvax — Measles virus vaccine (attenuate)administered subcutaneously at a single dose of 0.5 mL at 6 months of age
  Arms: 1
Biological: M-M-R-II — Measles-Mumps-Rubella vaccine (attenuated)administered subcutaneously as a single dose of 0.5 mL at 12 months of age

SUMMARY:
To compare measles seroconversion rates (development of antibodies) at 13 months of age in HIV-infected and uninfected children on one of two immunization schedules: attenuated measles/mumps/rubella virus (M-M-R II) vaccine at 12 months versus attenuated measles vaccine (Attenuvax) at 6 months plus M-M-R II vaccine at 12 months.

Recommendations for the age at vaccination should balance the need to minimize the risk of morbidity and mortality with the benefit of achieving the highest seroconversion rates. Immunizing a more intact immune system at an earlier stage of HIV infection may in turn achieve better and long-lasting measles protection. This study will help define a more effective measles vaccine regimen for children diagnosed with HIV infection and will provide greater insight into the functional status of the HIV-infected children's humoral immune system.

DETAILED DESCRIPTION:
Recommendations for the age at vaccination should balance the need to minimize the risk of morbidity and mortality with the benefit of achieving the highest seroconversion rates. Immunizing a more intact immune system at an earlier stage of HIV infection may in turn achieve better and long-lasting measles protection. This study will help define a more effective measles vaccine regimen for children diagnosed with HIV infection and will provide greater insight into the functional status of the HIV-infected children's humoral immune system.

Patients, HIV infected and uninfected, are randomized to one of two attenuated measles vaccine schedules: at 6 and 12 months of age, or at 12 months of age only. Attenuvax is administered as the month 6 vaccine and M-M-R II as the month 12 vaccine. Patients are followed for 24 months after the last vaccination.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Willing to have and receive results of HIV test
* Been born to mothers with HIV infection or history of AIDS-defining condition by CDC criteria.
* No history of opportunistic infection.
* No known exposure to measles within 14 days prior to study entry.
* CD4+ lymphocyte count >= 750 cells/mm3 or more than 15% at 6 months of age.
* Parent or legal guardian available to give written informed consent and be willing to comply with all study requirements.
* Childhood immunizations (other than measles) according to current recommendations of the Immunization Practice Advisory Committee and American Academy of Pediatrics.

NOTE:

* Coenrollment on other therapeutic protocols (except for ACTG 185) is permitted.

NOTE:

* Patients must be located in a geographical area where measles immunization at 12 months is standard of care.

Recommended:

* Childhood immunizations other than measles according to current guidelines.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Intercurrent illness and/or fever for 7 days.
* Known sensitivity or allergy to neomycin or eggs.

Concurrent Medication:

Excluded:

* IVIG.
* Uninterrupted or anticipated steroid therapy (>= 2 mg/kg/day) for more than 2 weeks duration.

Patients with the prior condition are excluded:

* Platelet count < 50,000/mm3 at any time prior to study entry.

Prior Medication:

Excluded:

* Any IgG preparation within the past 6 months.

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Comparison of measles seroconversion rates at 13 months of age between HIV-infected children vaccinated at 12 months of age and HIV-infected children vaccinated at 6 and 12 months of age | Throughout study
Comparison of seroconversion rates at 13 months of age (following second vaccination) of HIV-uninfected children with HIV-infected children. | Throughout study
Comparison of seroconversion rates at 13 months of age (following single vaccination) of HIV-uninfected children with HIV-infected children following vaccination at 12 months of age | Throughout study

SECONDARY OUTCOMES:
Comparison of measles seroconversion rates in HIV-infected children vaccinated at 6 months of age with HIV-infected children vaccinated at 12 months of age | Throughout study
Assessment of measles antibody decay and persistence in HIV-infected and HIV-unifected vaccinees | Throughout study
Evaluation of adverse effects and immune reactions to vaccine in HIV-infected children and HIV-uninfected vaccinees | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Chandwani S, Study Chair; Krasinski K, Study Chair
Locations (46):
- United States (43):
  - UAB, Dept. of Ped., Div. of Infectious Diseases, Birmingham, Alabama
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Emory Univ. School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Atlanta, Georgia
  - Cook County Hosp., Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Univ. of Illinois College of Medicine at Chicago, Dept. of Peds., Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - UMDNJ - Robert Wood Johnson, New Brunswick, New Jersey
  - NJ Med. School CRS, Newark, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey, Paterson, New Jersey
  - Children's Hospital at Albany Medical Center, Dept. of Peds., Albany, New York
  - North Shore-Long Island Jewish Health System, Dept. of Peds., Great Neck, New York
  - Schneider Children's Hosp., Div. of Infectious Diseases, New Hyde Park, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Metropolitan Hosp. Ctr., New York, New York
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - Med. Univ. of South Carolina, Div. of Ped. Infectious Diseases, Charleston, South Carolina
  - Texas Children's Hosp. CRS, Houston, Texas
  - Childrens Hosp. of the Kings Daughters, Norfolk, Virginia
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (3):
  - Univ. Hosp. Ramón Ruiz Arnau, Dept. of Peds., Bayamón
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan

REFERENCES:
- [Result] Chandwani S, Beeler J, Li H, Audet S, Smith B, Moye J, Nalin D, Krasinski K; PACTG 225 Study Team. Safety and immunogenicity of early measles vaccination in children born to HIV-infected mothers in the United States: results of Pediatric AIDS Clinical Trials Group (PACTG) protocol 225. J Infect Dis. 2011 Jul;204 Suppl 1(Suppl 1):S179-89. doi: 10.1093/infdis/jir089. PMID 21666159